CLINICAL TRIAL: NCT01229748
Title: Family Intervention for Teen Drinking and Alcohol-Related Crises in the ER
Brief Title: Family Intervention for Teen Drinking in the ER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Cynthia Rowe, Associate Professor, University of Miami
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 20090623
Record Dates: First submitted 2010-10-26; First posted 2010-10-28 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Multidimensional Family Therapy (Experimental): Multidimensional Family Therapy is an outpatient family-based treatment for troubled youth.(Liddle, 2002) considered in the U.S. and abroad as an empirically supported Best Practice treatment for teen substance abuse and delinquency (USDHHS 2002; Drug Strategies 2003; NIDA 1999; Rigter et al 2004).
  Interventions: Behavioral: Multidimensional Family Therapy
- Family Motivational Interviewing (Experimental): Motivational Interviewing (MI; Miller 1983; Miller & Rollnick 1991), is a client-centered treatment designed to strengthen clients' commitment and empower them to change their substance use behavior (Miller & Rollnick 2002).
  Interventions: Behavioral: Family Motivational Interviewing Intervention
- Standard Care (Other): The standard care condition will represent typical services for teens with alcohol problems in the community: assessment and referral for treatment
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Standard Care — Clients attend two 90-minute group sessions per week.Treatment lasts for three months.
  Arms: Standard Care
Behavioral: Multidimensional Family Therapy — Multidimensional Family Therapy is an outpatient family-based treatment for troubled youth (Liddle, 2002). Treatment duration is 3 months, sessions last 60-90 minutes, with an average of 2 sessions per week and additional extrafamilial work and phone contacts as needed.
  Arms: Multidimensional Family Therapy
Behavioral: Family Motivational Interviewing Intervention — Youth and parents receive 2 FMII sessions in their homes within 72 hours of the ER incident, and youth will be linked with group treatment lasting 3 months.
  Arms: Family Motivational Interviewing

SUMMARY:
The investigators propose a randomized controlled trial with five aims: 1. To investigate the engagement potential and effectiveness of a family-centered intervention (MDFT) and Family Motivational Interviewing Intervention (FMII)/group for teens with alcohol-related crises; 2. To explore differential treatment effects with comorbid adolescents; 3. To examine the role of motivation and family factors as treatment mediators; 4. To examine long-term abstinence, patterns and predictors of relapse up to 18 months follow-up; and 5. To compare the total and net monetary benefits to society of MDFT, FMII/group, and standard care.

DETAILED DESCRIPTION:
Aim 1: To investigate in a randomized controlled trial the engagement potential and effectiveness of family-centered intervention (MDFT) and family-involved MI (FMII) for teens with alcohol problems

* Hypothesis 1a: Treatment engagement will be higher in MDFT and FMII than in standard care as evidenced by higher numbers of MDFT and FMII youth enrolled in substance abuse treatment.
* Hypothesis 1b: Treatment completion will be higher for MDFT than FMII/group and standard care as evidenced by more teens/families in MDFT completing a full course of treatment.
* Hypothesis 1c: Youth assigned to MDFT and FMII/group will show greater decreases in alcohol use and binge drinking than youth in standard care at the 3 month follow-up (end of treatment). MDFT participants will show greater decreases in alcohol use and binge drinking than FMII/group and standard care during the post-treatment period and up to 18 month follow-up, and they will be less likely to meet diagnostic criteria for an AUD at 18 months.
* Hypothesis 1d: Youth assigned to MDFT and FMII/group will show greater reductions than youth in standard care in problems related to alcohol use, including drug use, drinking and driving, alcohol-related injury, health and mental health problems, school problems, delinquency, and association with substance abusing peers at the 3 month follow-up (end of treatment). Youth in MDFT will show greater reductions in these problems than FMII/group and standard care in the post-treatment period and up to 18 month follow-up.

Aim 2: To explore differential treatment effects with comorbid adolescents

* Hypothesis 2: For youth with low baseline levels of alcohol, drug, and psychiatric problems, MDFT and FMII/group will both be more effective than standard care. MDFT will reduce alcohol use more significantly than FMII/group for teens with more severe baseline alcohol, drug, and psychiatric problems.

Aim 3: To examine the contribution of motivation and family factors as mediators of treatment effects

* Hypothesis 3a: In both MDFT and FMII/group, motivation to change at the end of the initial engagement sessions in both teen and parent will predict treatment participation and 3 month outcomes (end of treatment) to a greater extent than motivation in the teen or parent alone.
* Hypothesis 3b: In both MDFT and FMII/group, effective parenting practices and strong family relationships will predict better alcohol and related outcomes at 3 month follow-up.

Aim 4: To examine long-term abstinence, patterns and predictors of relapse up to 18 months follow-up

* Hypothesis 4a: Four distinct patterns of relapse will emerge between 3 month and 18 month follow-up: high abstinence, low abstinence, decreasing abstinence, and increasing abstinence.
* Hypothesis 4b: MDFT youth will be more likely to be in the high abstinence and increasing abstinence groups; youth in FMII/group will be more likely to be in the decreasing abstinence group; and youth in standard care will be more likely to be in the low abstinence group.
* Hypothesis 4c: Youth in MDFT will show more significant reductions in risk factors for alcohol relapse (family dysfunction, lack of abstinence motivation, positive alcohol expectancies, poor abstinence coping, lack of support for abstinence) than youth in FMII/group or standard care.

Aim 5: To compare the total/net monetary benefits to society of MDFT, FMII/group, and standard care

* Hypothesis 5: MDFT and FMII/group will generate significantly higher total and net monetary benefits to society than youth in standard care at 18 months post-ER visit.
* Research Question 5: Will MDFT or FMII/group generate higher total/net benefits to society?

ELIGIBILITY:
Inclusion Criteria:

1. Between ages 12 to 18 years old
2. Present in ER/trauma unit
3. Meet minimum cut-off of 4 on the AUDIT; OR BAC of 0.01% or more on QED; OR report alcohol use within 6 hours of ER visit
4. Not receiving any other behavioral treatment
5. At least one parent/guardian is willing to participate in assessments and intervention
6. Parent consent/youth assent

Exclusion Criteria:

1. Meet DSM-IV dependence criteria for any substance other than alcohol, marijuana, or tobacco
2. Mental retardation or pervasive developmental disorders
3. Psychotic symptoms
4. Current suicidality

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2010-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Treatment engagement/retention | Proportion of adolescents enrolled in substance abuse treatment at 3 months post -intake.
  To investigate the engagement potential and effectiveness of a family-centered intervention (MDFT) and family-involved MI (FMII) for teens with alcohol-related crises.

SECONDARY OUTCOMES:
Alcohol use/abstinence | Youth assigned to MDFT and FMII/group will show greater decreases in alcohol use and binge drinking than youth in standard care at 3 months post intake.
  MDFT participants will show greater decreases in alcohol use and binge drinking than FMII/group and standard care during the post-treatment period and up to 18 month follow-up, and they will be less likely to meet diagnostic criteria for an AUD at 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia L Rowe, PhD, Principal Investigator — University of Miami
Locations (3):
- United States (3):
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Miami Children's Hospital, Miami, Florida

REFERENCES:
- [Background] Rowe CL, Liddle HA. Family-based treatment development for adolescent alcohol abuse. Int J Adolesc Med Health. 2006 Jan-Mar;18(1):43-51. doi: 10.1515/ijamh.2006.18.1.43. PMID 16639858